CLINICAL TRIAL: NCT00182377
Title: A Randomized, Prospective, Blinded Clinical Trial to Evaluate the Efficacy and Safety of Pentastarch Use in Patients Undergoing Coronary Artery Bypass Surgery or Valve Replacement Surgery Using Cardiopulmonary Bypass Circuits
Brief Title: Pentastarch Use in Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 02-183
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2004-09

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
Keywords: patients undergoing cardiac surgery requiring cardiopulmonary bypass
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

INTERVENTIONS:
Drug: Pentastarch (displace either 500 ml or 1000 ml of pump prime with pentastarch)

SUMMARY:
Patients undergoing cardiac surgery with cardiopulmonary bypass require significant fluid administration. Fluids are used routinely to replace blood lost during and after surgery. Significant amounts of fluid are also used to prime the tubing and components of the cardiopulmonary bypass pump before and during its use. The use of Pentaspan - a synthetic pentastarch - was started because of the restriction of use for blood and blood products, particularly albumin. Pentaspan is usually used after surgery in the Intensive Care Unit (ICU). The impact of the use of pentastarch on coagulation, fluid balance and bleeding are very limited. This study will methodically evaluate the impact of using increasingly greater amounts of pentastarch during surgery on an open heart surgery patient's recovery in particular - is there more bleeding, does his/her blood clot as well, and how much fluid overall is used and excreted?

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing either coronary artery bypass surgery or valve surgery requiring the use of cardiopulmonary bypass circuit

Exclusion Criteria:

* Emergency surgery
* Regurgitant valve pathology
* Redo surgery
* Significant left ventricular (LV) dysfunction
* Significant renal insufficiency
* Anticipation of associated procedure - eg carotid endarterectomy
* Ongoing sepsis or endocarditis
* Received aspirin (ASA) or Plavix within 96 hours of surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
transfusion requirements
fluid balance

SECONDARY OUTCOMES:
postoperative bleeding
mediastinal drainage
coagulation parameters
respiratory status

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cybulsky, MD, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - General Division, Hamilton, Ontario, Canada